CLINICAL TRIAL: NCT06423352
Title: A Phase 1/2, Randomized, Double-blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacodynamics, and Pharmacokinetics of Zilebesiran in Japanese Patients With Mild to Moderate Hypertension
Brief Title: A Study to Evaluate Zilebesiran in Japanese Patients With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALN-AGT01-006
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Mild to Moderate Hypertension
Keywords: High blood pressure; Hypertension; Hypertensive; siRNA; Angiotensinogen; AGT
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Zilebesiran (Experimental): Participants will be administered a single dose of zilebesiran.
  Interventions: Drug: Zilebesiran
- Placebo (Placebo Comparator): Participants will be administered a single dose of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zilebesiran — Zilebesiran administered by subcutaneous (SC) injection
  Other Names: ALN-AGT01
  Arms: Zilebesiran
Drug: Placebo — Placebo administered by SC injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, efficacy, pharmacodynamics (PD) and pharmacokinetics (PK) of zilebesiran in Japanese patients with mild to moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Must have been born in Japan, and their biological parents and grandparents must have been of Japanese origin
* Has mean systolic office blood pressure (SBP) of >130 and <=165 mmHg by automated office blood pressure measurement, after a minimum of 3 weeks of washout if taking hypertensive medication
* Has 24-hour mean SBP ≥130 mmHg by ambulatory blood pressure monitoring (ABPM), without antihypertensive medication

Exclusion Criteria:

* Has secondary hypertension, symptomatic orthostatic hypotension
* Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2× upper limit of normal (ULN)
* Has elevated serum potassium >5 mmol/L
* Has estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73m^2
* Has received an investigational agent within the last 30 days
* Has Type 1 diabetes mellitus, poorly controlled Type 2 diabetes mellitus or newly diagnosed Type 2 diabetes mellitus
* Has history of intolerance to SC injection(s)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) | Up to 12 months

SECONDARY OUTCOMES:
Percent Change from Baseline in Serum Angiotensinogen (AGT) at Month 3 and Month 6 | Baseline and Month 3 and Month 6
Change from Baseline at Month 3 and Month 6 in 24-hour Mean Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Assessed by Ambulatory Blood Pressure Monitoring (ABPM) | Baseline and Month 3 and Month 6
Change from Baseline at Month 3 and Month 6 in SBP and DBP Assessed by Office Blood Pressure | Baseline and Month 3 and Month 6
Pharmacokinetics of Zilebesiran and its Metabolite assessed by Plasma Concentration | Predose and up to 3 days postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (3):
- Japan (3):
  - Clinical Trial Site, Fukuoka
  - Clinical Trial Site, Osaka
  - Clinical Trial Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Access to data may be declined where there is likelihood a patient could be identified or other feasibility issue, where there is a potential conflict of interest, a planned business activities or an actual or potential competitive risk. Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Timeframes for data access may vary and can take up to 6 months or more.
  Requests for access to data can be submitted via the website www.vivli.org. Questions can also be directed to datasharing@alnylam.com.